CLINICAL TRIAL: NCT00871455
Title: Effect of Low-Dose Baclofen Administration on the GH-IGF1 Axis Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4162C-7
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Baclofen; Growth Hormone, Pituitary; Insulin-Like Growth Factor I
MeSH Terms: conditions — Spinal Cord Injuries; Pituitary Diseases | interventions — Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Subjects will receive 20 mg baclofen for 8 weeks, followed by 40 mg baclofen for 8 weeks.
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Baclofen — Subjects will receive 20 mg baclofen for 8 weeks, followed by 40 mg baclofen for 8 weeks.

SUMMARY:
Insulin-like growth factor I (IGF-I) is used as a measure of the body's ability to produce growth hormone. Growth hormone is important for muscle tissue as well as many other tissues in the body. Growth hormone (GH) and IGF-I have been shown to be reduced in many persons with SCI. Baclofen is a FDA approved drug that is used to treat spasticity. Persons receiving long-term baclofen therapy have been demonstrated to have increased growth hormone and IGF-I levels. IGF-I levels will be determined before and after treatment with baclofen. In this study, the investigators will determine the minimum dose of baclofen at which improvements in GH and IGF-1 levels occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic SCI (injury greater than 6 months) who have been screened and found to have depressed plasma IGF-1 levels and who are not taking baclofen.

Exclusion Criteria:

* Acute illness of any etiology,
* Patients with chronic renal, liver, lung, or cardiac disease,
* Patients receiving any of the following medications: narcotics, or L-DOPA, and
* Alcoholics.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-04; Primary Completion 2007-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Determine the threshold dose 20 or 40 mg/d of baclofen and the dose-response curve of the medication for its effect to raise plasma IGF-1 levels | 20-week (5 months) in which subjects are asked to report for 12 visits after starting baclofen therapy

SECONDARY OUTCOMES:
Assessment of the adverse side effects, if any, of low dose baclofen therapy | 20-week (5 months) in which subjects are asked to report for 12 visits after starting baclofen therapy

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States